CLINICAL TRIAL: NCT06881212
Title: Effects Of Therapeutic Approaches On Intubation Response, Agitation Behavior, And Extubation Time İn Patients Undergoing Open Heart Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Nareg Dogan, Associate Prof, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E-54022451-050.05.04-73654
Record Dates: First submitted 2025-01-22; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Cardiac Surgery Subjects; Nursing Care
Keywords: Education,; Nursing; Cardiovascular Surgery; Therapeutic Approach

STUDY DESIGN:
Intervention Model Description: The research is a quasi-experimental study with a post-test experimental-control group.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Trained group (Experimental): Pre-Surgery:
  Patients received a special training including therapeutic communication techniques.
  The training was prepared by reviewing the literature and integrated into hospital practices.
  One day before surgery, the patient and patient's relatives were trained in a session lasting 40-50 minutes.
  All stages of the training were monitored using the "Preoperative Training Checklist ".
  Postoperative:
  When the patients were taken to the intensive care unit, sedation was applied again at the first awakening according to the hospital protocol.
  After the effect of sedation wore off and the patient was conscious but still intubated, therapeutic interventions were performed.
  This process was done with the "Postoperative Education Checklist " prepared based on the literature.
  Data Collection:
  4 hours after the patients woke up, by the researcher: RASS (Richmond Agitation Sedation Scale) was applied. Intubation Reactions Form was filled. The time to come out of intubation was recorded.
  Interventions: Behavioral: THERAPEUTIC APPROACH TRAINING
- Non-training group (No Intervention): Preoperative No special training was given to the control group. Patients were only subjected to routine hospital procedures.
  Postoperative:
  Standard hospital protocol was applied when the patients were admitted to the intensive care unit.
  Sedation was applied again, but no additional therapeutic intervention was performed.
  Patients received only routine nursing care.
  Data Collection:
  4 hours after patients woke up, by the investigator: RASS (Richmond Agitation Sedation Scale) was administered. Intubation Reactions Form was completed. The time to come out of intubation was recorded.

INTERVENTIONS:
Behavioral: THERAPEUTIC APPROACH TRAINING — This study focuses on pre- and post-operative training for open-heart surgery patients, aiming to reduce anxiety, agitation, and discomfort during intubation and recovery.
  In the meeting phase, the nurse introduces herself, explains the research, and obtains written/verbal consent. The patient's anxiety level is assessed.
  In the study phase, patients are informed about the surgical process, breathing exercises, Intensive Care Unit conditions, and postoperative care. They are encouraged to express fears and concerns to improve psychological preparedness.
  Key topics include:
  Fasting before surgery Breathing exercises to ease extubation Use of mechanical ventilation Intensive Care Unit environment & pain management Early mobilization & recovery timeline Patients receive guidance on their role in recovery, ensuring better adaptation and reduced distress post-surgery.
  Arms: Trained group

SUMMARY:
This study was conducted to understand how training given to patients before and after open-heart surgery affects their reactions during intubation (when a breathing tube is inserted), their agitation levels, and the time it takes to remove the breathing tube.

Study Design

The research followed a quasi-experimental design, meaning patients were divided into two groups:

Experimental Group - Received special training before and after surgery. Control Group - Received standard hospital care without additional training. Key Variables Independent Variable (What was changed): The training given before and after surgery.

Dependent Variables (What was measured):

Patient reactions during intubation Agitation levels Time taken to remove the breathing tube Study Hypotheses Patients who received the training would show different reactions compared to those who did not.

1.1. The trained group would show fewer negative reactions during intubation. Patients who received the training would have different agitation levels compared to the control group.

2.1. The trained group would be less agitated. The time taken to remove the breathing tube would be different between the two groups.

3.1. The trained group would have their breathing tube removed faster. Where and When Was the Study Conducted? The research took place at Bezmialem Vakif University Hospital in Istanbul in the cardiovascular surgery department, between October 10, 2022 - January 7, 2023.

Participants The study initially considered 123 patients who had undergone open-heart surgery during this period.

Patients were selected based on certain health conditions and criteria (age, no chronic respiratory disease, type of surgery, etc.).

After applying these criteria, 30 patients (15 in each group) were included in the final study.

How Were Patients Selected? To ensure fairness, patients were randomly assigned to either the experimental or control group.

A computer-generated random list was used to assign them. Who Was Included in the Study? Patients who had Coronary Artery Bypass (CABG), Aortic Valve Replacement (AVR), or Mitral Valve Replacement (MVR) surgery.

Patients aged 45-70 years old. Who Was Excluded? Patients with chronic respiratory disease (as it could affect intubation time). Patients who had previous open-heart surgery (as prior experience could influence their reaction).

Patients who did not speak Turkish or had cognitive issues. Patients with severe psychiatric conditions. Data Collection & Training Process

Before the surgery:

Patients were asked about their age, gender, smoking habits, medical history, and other factors.

Their anxiety levels were measured using a scale from 0 to 10 (0 = No anxiety, 10 = Extreme anxiety).

Training for the experimental group:

A special 40-50 minute training session was given a day before surgery. The training included breathing techniques, relaxation methods, and information about what to expect during recovery.

Family members were also involved.

After the surgery:

Patients were sedated as part of hospital protocol and then observed when they first woke up in the Intensive Care Unit (ICU).

The trained group received additional therapeutic communication techniques when they first woke up to help them stay calm.

The control group received only standard hospital care. Four hours after waking up, all patients were evaluated for their agitation levels and reactions to intubation.

How Were Reactions Measured? Richmond Agitation Sedation Scale (RASS ) - This measured how restless or calm the patient was.

Observation of Intubation Reactions - The research team noted behaviors such as:

Trying to pull out the breathing tube Biting the tube Facial expressions (like frowning or grimacing) Grabbing bed sheets Moving legs restlessly Breathing in sync with the ventilator Each behavior was scored from 0 (Not observed) to 4 (Strongly observed). A higher score meant the patient was more uncomfortable with intubation.

Results General reactions to intubation (measured with a scale) were similar in both groups.

However, when specific behaviors were examined, the control group had more visible distress:

More frowning and wrinkled facial expressions (p=0.030). More grabbing of bed sheets (p=0.013). There was no significant difference in agitation levels between the two groups. The time taken to remove the breathing tube was also not significantly different between the two groups.

Conclusion The special pre- and post-surgery training helped patients remain more comfortable during intubation, reducing visible signs of distress.

However, the training did not significantly impact overall agitation levels or the time needed to remove the breathing tube.

This suggests that therapeutic communication techniques may improve patient comfort but do not necessarily speed up the recovery process.

ELIGIBILITY:
Inclusion Criteria:

* Coronary Artery Bypass Graft, Aortic Valve Replacement, Mitral Valve Replacement having undergone one of these operations
* No Chronic Respiratory Disease

Exclusion Criteria:

* Aortic Valve Replacement and Mitral Valve Replacement performed together
* Use of a method other than median sternotomy
* Redo coronary bypass surgery
* Illiteracy and not knowing Turkish
* Being under psychiatric treatment and follow-up recently (last 1 year)

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2023-01-07 (Actual); Study Completion 2023-01-07 (Actual)

PRIMARY OUTCOMES:
Sociodemographic information form | From the data obtained from the enrollment of the first participant until week 12 Before the operation
  The demographic characteristics of the patients such as age, gender, education level, chronic diseases, history of surgery, height and weight, smoking and alcohol use, psychiatric treatment and follow-up status were evaluated with a 13-item form created by the researchers by using the literature.
Numerical anxiety scale | From the data obtained from the enrollment of the first participant until week 12 Before the operation
  The Numerical Anxiety scale has a starting point of "0" or "no anxiety" and an ending point of '10' or "severe anxiety" (horizontal line was used in this study). The patient chooses the number from the scale that best describes him/her. Preoperative and postoperative anxiety is higher in patients undergoing open heart surgery compared to other surgeries. Anxiety level is a factor that may lead to increased agitation and patient non-compliance with mechanical ventilator. For this reason, anxiety level was used as a control variable to measure the effectiveness of the intervention to be applied to the experimental and control groups and to ensure the homogeneity of the experimental and control groups. The results of the scale were evaluated on the arithmetic mean.

OTHER OUTCOMES:
Richmond Agitation Sedation Scale (RASS) | Within 12 weeks after the initial registration date,after the operation
  The scale was developed by the Virginia Commonwealth University of Richmond. In the scale, which has a total score of 10, the patient's agitation is scored in the reference range of +4 (combative; potentially dangerous for staff) to -5 (cannot be aroused). Scoring is done as; +4 belligerent, +3 very agitated, +2 agitated, +1 restless, 0 calm/awake, -1 sleepy, -2 light sedation, -3 moderate sedation, -4 deep sedation and -5 coma. A positive score indicates that the patient is agitated and a negative score indicates that the patient is in a coma or under the influence of sedation .Written permission for the scale was obtained via e-mail.
Intubation responses observation form | Within 12 weeks after the initial registration date after the operation
  In this observation form, 6 of the most common behaviors (Trying to pull the intubation tube, biting the intubation tube, wrinkled facial expression, collecting sheets with hands, trying to take the legs out of the bed railing, showing compliance with the ventilator) were examined by examining the literature and taking into account the changes indicated by 8 experts in the field according to the opinion form. In the form consisting of 6 sections, each item is graded on a 5-point Likert-type scale. (0=Behavior Not Observed; 4=Sustained Observed) The intubation behaviors observation form score is obtained by summing the scores of the questions. A high score indicates poor compliance with intubation. The Cronbach's alpha value of this scale was determined as 0.824 for this study.Intubation length of stay was recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Gedik University, Istanbul, Kartal, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
I WANT TO PUBLISH IT AS AN ARTICLE IN A SCIE INDEXED JOURNAL
Supporting Information: Study Protocol, SAP, CSR, Analytic Code

REFERENCES:
- [Background] Tully PJ, Baker RA. Depression, anxiety, and cardiac morbidity outcomes after coronary artery bypass surgery: a contemporary and practical review. J Geriatr Cardiol. 2012 Jun;9(2):197-208. doi: 10.3724/SP.J.1263.2011.12221. PMID 22916068
- [Background] Hoyer J, Eifert GH, Einsle F, Zimmermann K, Krauss S, Knaut M, Matschke K, Kollner V. Heart-focused anxiety before and after cardiac surgery. J Psychosom Res. 2008 Mar;64(3):291-7. doi: 10.1016/j.jpsychores.2007.09.009. PMID 18291244
- [Background] İnce, F. (2020). Kardiyak cerrahi öncesi uygulanan eğitimin anksiyete, depresyon, yaşam kalitesi ve kinezyofobi üzerine etkisi (Master's thesis, İstanbul Medipol Üniversitesi Sağlık Bilimleri Enstitüsü).
- See also: Calculatorsoup.com. Random Number Generator. (2022) (Accessed: 16.08.2022). — https://www.calculatorsoup.com/calculators/statistics/random-number-generator.php